CLINICAL TRIAL: NCT02941536
Title: Prospective Evaluation of Correlation Between Circulating Tumor Cells and Brain Disease Control After Focal Stereotactic Radiotherapy for Encephalic Metastases of Breast Cancer
Brief Title: Correlation Between Circulating Tumor Cells and Brain Disease Control After Focal Radiotherapy for Metastases of Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AC Camargo Cancer Center (Other)
Collaborators: International Atomic Energy Agency (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2258/16
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Brain Cancer; Breast Cancer
Keywords: Circulating Tumor Cells; Stereotactic Radiosurgery
MeSH Terms: conditions — Brain Neoplasms; Breast Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Circulating Tumor Cells and Radiotherapy (Other): Circulating tumor cells evaluation before and 4-5 weeks after focal stereotactic radiotherapy in single (SRS) or fractionated (SFRT) dose and correlate with the local and distant brain progression free survival in patients with metastatic breast cancer
  Interventions: Diagnostic Test: Circulating tumor cells evaluation

INTERVENTIONS:
Diagnostic Test: Circulating tumor cells evaluation — Sample collection of circulating tumor cells (CTC) before and 4-5 weeks after focal stereotactic radiotherapy in single (SRS) or fractionated (SFRT) dose.

SUMMARY:
This study assesses the number of CTCs before and 4-5 weeks after focal stereotactic radiotherapy, in single or fractionated dose, and correlate with the local and distant brain progression-free survival in patients with metastatic breast cancer.

DETAILED DESCRIPTION:
Brain metastases (BM) are the most prevalent tumors of the central nervous system (CNS), with a ratio of 10: 1 relative to primary tumors. In breast cancer, BM are becoming more frequent due to longer life expectancy. Patients with HER2-positive metastatic disease are prone to develop BM more often and they occur in 20 - 40% of cases. Circulating tumor cells (CTC) originate from the primary tumor and can migrate to distant organs. The possible correlation between CTC and the incidence of brain metastases could help define radiotherapy in patients with oligometastatic or not so widespread disease in the brain. However, there are few studies that evaluate these scenarios. Purpose: To assess the number of CTC before and 4-5 weeks after focal stereotactic radiotherapy in single (SRS) or fractionated (SFRT) dose and correlate with the local and distant brain progression free survival in patients with metastatic breast cancer. Potential invasion markers in these cells will be evaluated and correlated with clinical outcome. Patients and Methods: Prospective, single-center research which will be developed at the Radiation Oncology Department of AC Camargo Cancer Center. Patients with diagnosis of metastatic breast cancer to the brain with an indication of focal radiotherapy, SRS or SFRT, will be recruited. The blood will be collected and processed for analysis of CTC by the ISET method (Rarecells, France). The invasion markers (HER-2, COX-2, EGFR, Notch 1 and ST6GALNAC5) will be analyzed on CTC by immunocytochemistry. Expected Results: If our hypothesis is proven, we may include the analysis and quantification of CTC in clinical practice as early indicator of local or distant recurrence in the brain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of BM of breast cancer and indication of focal radiotherapy to the brain lesions.

Exclusion Criteria:

* Patients who received WBRT less than 30 days from the initial CTC dosage.
* Patients who received systemic treatment for less than 7 days of the initial CTC dosage.
* Pregnant patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Brain progression-free survival | 6 months
  Local and Distant brain progression

SECONDARY OUTCOMES:
Overall survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Douglas G Castro, MD, MSc, Principal Investigator — AC Camargo Cancer Center
Locations (1):
- AC Camargo Cancer Center, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: 6 months after article publication
Access Criteria: Correlated Area Investigators with publishing background and a defined objective.